CLINICAL TRIAL: NCT07038187
Title: Effect of Music on Anxiety Levels During Intrauterine Device Application: A Randomized Controlled Trial
Brief Title: Effect of Music on Anxiety Levels During Intrauterine Device Application
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Şükriye ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, Şükriye ŞAHİN, Research Assistant Doctor, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025/0101
Record Dates: First submitted 2025-05-06; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Family Planning; Music Intervention
Keywords: THERAPY; FAMİLY PLANNİNG; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening with Binaural Beats (Experimental): Participants in the experimental group will listen to instrumental music embedded with 7 Hz binaural beats (theta range) generated using Gnaural (GPL-2.0 licensed, programmable sound generator). The tracks include piano and instrumental music played at a volume of 50-60 dB, allowing communication with the healthcare provider. Music will be delivered via headphones for approximately 30 minutes (20 minutes before and during the procedure). STAI-I and STAI-II scores will be assessed pre- and post-procedure.
  Interventions: Behavioral: Music Listening (Binaural Beats via Gnaural)
- Routine Care Without Music (No Intervention): Participants in the control group will receive standard care during IUD insertion. No music or other additional intervention will be applied. STAI-I and STAI-II scores will be measured before and after the procedure.

INTERVENTIONS:
Behavioral: Music Listening (Binaural Beats via Gnaural) — Modern 'relaxation' music regularly includes binaural beats. Binaural beats can be defined as a sensation produced by the arrival of sine tones of different frequencies in each ear. This sensation is created by the difference in frequency between the two tones reaching the ear. Music with binaural beats has been associated with reduced anxiety and increased relaxation by activating theta and delta wavelengths in the electroencephalography (EEG). The authors used Gnaural (GPL-2.0), a freely programmable sound generator, for the binaural beats. Two pieces of instrumental 7 Hz binaural beats were used, a piano and an instrumental. The music volume was between 50-60 decibels and was at a level where the participant could hear the healthcare professional performing the procedure.
  Arms: Music Listening with Binaural Beats

SUMMARY:
This study was conducted as a pre-test/post-test, randomized controlled trial to evaluate the effect of music on anxiety levels of women undergoing intrauterine device (IUD) insertion. Data were collected between January 2025 and May 2025 at a Community Health Center in Bingöl province. A total of 60 women (30 in the experimental group, 30 in the control group) who applied for IUD insertion were included. Women in the experimental group listened to slow classical music (12-15 beats per minute) through headphones for approximately 20 minutes prior to the procedure and continued listening during the procedure, totaling 30 minutes. Women in the control group did not listen to music. Anxiety levels were assessed before and after the procedure using the State-Trait Anxiety Inventory-State (STAI-S) Scale. Institutional and ethics committee approvals, as well as informed consent, were obtained before the study.

DETAILED DESCRIPTION:
This randomized controlled study aimed to assess the effect of music on procedural anxiety in women undergoing IUD insertion. Randomization was performed using a computer-generated random number table prepared by a statistician. Each participant meeting the inclusion criteria was assigned to either the experimental or control group via opaque envelopes distributed in the order of clinic admission. The independent variable was music listening, and the dependent variable was anxiety level measured using the STAI-S Scale. Data were collected from women at a Community Health Center between January and May 2025. The study received ethical approval and informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Women who will have an IUD for the first time
* Women aged 18-45

Exclusion Criteria:

* Women with hearing problems
* Women with psychiatric diagnoses

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants were included in the study because intrauterine device (IUD) was used as a family planning method.
Enrollment: 60 (Actual)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Anxiety severity | Baseline (immediately before the IUD procedure) and Post-Procedure (within 30 minutes after the IUD procedure)
  Anxiety severity will be measured using the State Anxiety subscale of the Spielberger State-Trait Anxiety Inventory (STAI-S). Participants will respond to 20 items using a 4-point Likert scale (1 = Not at all, 2 = Somewhat, 3 = Moderately so, 4 = Very much so).

SECONDARY OUTCOMES:
Trait Anxiety Severity | Baseline (immediately before the IUD procedure) and Post-Procedure (within 30 minutes after the IUD procedure)
  Trait anxiety will be measured using the Trait Anxiety subscale of the Spielberger State-Trait Anxiety Inventory (STAI-T), consisting of 20 items rated on a 4-point Likert scale. This scale assesses the participant's general tendency toward anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şükriye Şahin, PhD, Study Director — Kocaeli University; Yasemin Özhanlı, Assistant Professor, Study Chair — Kocaeli University; Elif Ayfer Baltacı Yıldız, PhD, Study Chair — Bingol University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No